CLINICAL TRIAL: NCT00495027
Title: Brief Cognitive-Behavioral Treatment for Victims of Mass Violence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH066589-02 (NIH)
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Last update posted 2007-07-02 (Estimated); Status verified 2007-06

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; prevention; World Wide Web; Behavior Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Internet-delivered Stress Innoculation Training

SUMMARY:
The objective of this randomized control trial is to compare the effectiveness of Stress Inoculation Training (SIT), a well researched psychological treatment for Post Traumatic Stress Disorder (PTSD), to that of the non-specific standard care provided in primary care settings, called Supportive Counseling (SC), on individuals who were exposed to the September 11, 2001 terrorist attack on the Pentagon, or the immediate aftermath of this attack. Both SIT and SC interventions will each be provided in one 2-hour session with eight weeks of daily systematic web-based follow up to promote self-help. The primary hypothesis of this study is that SIT will reduce the level of PTSD in participants relative to SCand to the pre-treatment levels.

DETAILED DESCRIPTION:
Because resources are often scarce in the aftermath of disasters, a useful mental health intervention is one that is effective, feasible, rapidly available, and efficiently delivered to the largest proportion of affected individuals possible. In terms of treating PTSD in other trauma contexts, there is considerable evidence that cognitive-behavioral therapy (CBT) procedures are effective at reducing the array of PTSD symptoms. Overall, the available evidence points to the theoretical and empirical justification for using Prolonged Exposure (PE) and Stress Inoculation Training (SIT), two components of CBT, with patients presenting with PTSD. A practical limitation of available studies is that they are limited to individually administered therapy contexts that typically require between 8 and 12 sessions delivered in a specialty mental health care-setting. The labor-intensive nature of these therapies represents a significant obstacle to provision of therapy to potentially thousands of individuals suffering PTSD in the context of mass violence events.

The major aim of this project is to evaluate an abbreviated format of SIT that aims to provide effective self/stress-management skills to individuals with PTSD. The rationale behind this intervention is that with appropriate and intensive therapist input during a single session of therapy, supplemented systematically with self-paced and self-directed homework, promoted, prompted, and monitored via a specialized web-site and augmented by therapist feedback and guidance delivered via the web, primary care patients with PTSD stemming from mass violence can benefit from the strategies that have demonstrated efficacy in reducing PTSD symptoms. Survivors of the Pentagon attack on 9/11 who present at primary care clinics that serve the Pengaton are randomly assigned to SIT or a supportive counseling control group. Patients' compliance and symptoms are monitored on the web and via clinical interview.

ELIGIBILITY:
Inclusion Criteria:

1. Sufficient proximity to the September 11, 2001 Pentagon attack and its aftermath, including rescue and clean-up activities (at least two items endorsed on the exposure checklist, see the checklist on page 6 of the attached Rapid protocol)
2. At least one re-experiencing symptom rated as "severe" on the Post Traumatic Stress Disorder Checklist (PCL)

Exclusion Criteria:

1. Substance dependent
2. Current suicidal ideation
3. History of psychotic disorder
4. Inadequate comprehension of English
5. Evidence of PTSD or depression immediately prior to the attack
6. Currently receiving psychological/psychiatric treatment.
7. Marked dissociative presentation.
8. Grossly inadequate social supports
9. Mental retardation and cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2002-03; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
PTSD Symptom Scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Brett T Litz, Ph.D., Principal Investigator — Boston University
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States